CLINICAL TRIAL: NCT01799083
Title: Phase 1/2 Study of Decitabine Alone and/or in Combination With Chemotherapy and/or Cytokine Induced Killer Cell Transfusion in Patients With Relapsed or Refractory Solid Tumors and B Cell Lymphomas
Brief Title: Lower Dose Decitabine Based Therapy in Patients With Refractory and/or Chemotherapy Resistant Solid Tumors or B Cell Lymphomas
Acronym: CIK
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Han weidong (Other)
Responsible Party: Sponsor-Investigator, Han weidong, Researcher, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-002
Record Dates: First submitted 2013-02-22; First posted 2013-02-26 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Solid Tumors; B Cell Lymphoma
Keywords: Advanced solid tumors; B cell lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Decitabine (Experimental): A continuous 5-day treatment of lower dose decitabine within 4-6 weeks is regarded as a treatment cycle, transfusion of auto-CIK cells or chemotherapy regimen may be used for patients.
  Interventions: Drug: Decitabine; Biological: cytokine-induced killer cell

INTERVENTIONS:
Drug: Decitabine — A continuous 5-day lower-dose decitabine transfusion will be performed for patients during each treatment cycle, and autologous cytokine-induced killer cells may be transfused or chemotherapy may be also added.
  Other Names: Dacogen
Biological: cytokine-induced killer cell — Autologous cytokine-induced killer cells may be used for patients before and after decitabine treatment.
  Other Names: CIK transfusion

SUMMARY:
Determine alone or in combination with chemotherapy or autologous cytokine induced killer cells are effective and safe in the treatment of patients with relapsed and/or refractory solid tumors or B Cell lymphomas.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether lower dose decitabine based therapy is safe and can effectively control tumor progression.

ELIGIBILITY:
Inclusion Criteria:

* Solid Tumor

  * Histologically confirmed advanced solid tumor
  * 1 to 3 prior treatment regimens
  * At least one site of radiographically measurable disease of ≥ 2 cm in the largest dimension by traditional computerized tomography (CT) scanning technique or ≥ 1 cm in the largest dimension by spiral CT scanning (per RECIST criteria); or if, in the Principal Investigator's opinion, evaluable disease can be reliably and consistently followed, the subject may be eligible upon approval by the Medical Monitor
* B Cell Lymphoma

  * Histologically or cytologically confirmed B Cell Lymphoma.
  * Patients must have had an initial diagnosis of B Cell NHL (including follicular, small lymphocytic, lymphoplasmacytoid, and marginal zone lymphoma), indolent disease that transformed to a more aggressive subtype, as previously described or patients may have mantle cell lymphoma.
  * Patients are required to have received prior chemotherapy (alone or combined with rituximab or other treatment) and are considered refractory to (defined as no response, or progression within 6 months of completing therapy) or intolerant of continued rituximab or other treatment.
  * Patients may have received up to a maximum of four prior unique chemotherapy regimens, including if not contra-indicated autologous stem-cell transplantation (ASCT).
  * For patients to enroll in the expanded dose group for lymphoma, patients must have measurable disease

Exclusion Criteria:

* Disease Related

  * Chemotherapy with approved or investigational anticancer therapeutics, including steroid therapy, within 3 weeks prior to first dose or 6 weeks for antibody therapy
  * Radiation therapy or immunotherapy within 3 weeks prior to first dose (except for antibody therapy, where 6 weeks is required); localized radiation therapy within 1 week prior to first dose
  * Subjects with prior brain metastases are permitted, but must have completed treatment and have no evidence of active central nervous system (CNS) disease for at least 4 weeks prior to first dose
  * For lymphoma patients; patients with prior stem cell transplant therapy (autologous SCT within the prior 8 weeks; allogeneic SCT within the prior 16 weeks). Patients with prior allogeneic SCT should not have evidence of moderate-to-severe GVHD.
  * Participation in an investigational therapeutic study within 3 weeks prior to first dose
  * Prior treatment with decitabine

Concurrent Conditions

* Major surgery within 3 weeks prior to first dose
* Congestive heart failure (New York Heart Association class III to IV), symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention, or myocardial infarction within 3 months prior to first dose
* Acute active infection requiring systemic antibiotics, antivirals, or antifungals within 2 weeks prior to first dose
* Known or suspected HIV infection or subjects who are HIV seropositive
* Active hepatitis A, B, or C infection
* Significant neuropathy (Grade 3, Grade 4, or Grade 2 with pain) at the time of the first dose

Ethical / Other

* Female subjects who are pregnant or lactating
* Any clinically significant psychiatric or medical condition that in the opinion of the Investigator could interfere with protocol adherence or a subject's ability to give informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Response confirmed by non-investigational CT or MRI, or confirmed by biopsy | within the first 30 days after four-cycle treatment

SECONDARY OUTCOMES:
tumor marker | at least once within 30 days afther completing four-cycle treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Biotherapeutic Department of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Lu XC, Yang B, Yu RL, Chi XH, Tuo S, Tuo CW, Zhu HL, Wang Y, Jiang CG, Fu XB, Yang Y, Liu Y, Yao SQ, Dai HR, Cai L, Li BJ, Han WD. Clinical study of autologous cytokine-induced killer cells for the treatment of elderly patients with diffuse large B-cell lymphoma. Cell Biochem Biophys. 2012 Jan;62(1):257-65. doi: 10.1007/s12013-011-9273-6. PMID 21913005
- [Background] Yang B, Lu XC, Yu RL, Chi XH, Liu Y, Wang Y, Dai HR, Zhu HL, Cai LL, Han WD. Repeated transfusions of autologous cytokine-induced killer cells for treatment of haematological malignancies in elderly patients: a pilot clinical trial. Hematol Oncol. 2012 Sep;30(3):115-22. doi: 10.1002/hon.1012. Epub 2011 Aug 23. PMID 22972689
- [Derived] Fan H, Lu X, Wang X, Liu Y, Guo B, Zhang Y, Zhang W, Nie J, Feng K, Chen M, Zhang Y, Wang Y, Shi F, Fu X, Zhu H, Han W. Low-dose decitabine-based chemoimmunotherapy for patients with refractory advanced solid tumors: a phase I/II report. J Immunol Res. 2014;2014:371087. doi: 10.1155/2014/371087. Epub 2014 May 21. PMID 24963497
- [Derived] Zhang Y, Wang J, Wang Y, Lu XC, Fan H, Liu Y, Zhang Y, Feng KC, Zhang WY, Chen MX, Fu X, Han WD. Autologous CIK cell immunotherapy in patients with renal cell carcinoma after radical nephrectomy. Clin Dev Immunol. 2013;2013:195691. doi: 10.1155/2013/195691. Epub 2013 Dec 9. PMID 24382970